CLINICAL TRIAL: NCT03854916
Title: Caminamos: A Location-based Smartphone App for Latinas to Connect With Nearby Walking Partners Ph II
Brief Title: Caminamos: A Smartphone App for Latinas to Connect With Walking Partners
Acronym: Caminemos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0321; R44MD009652-02 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2019-02-26 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Physical Activity
Keywords: Physical Activity; Latina; Hispanic; Women; Minority Health; Mobile Technology; Social Support; mHealth; Location-based Services; Walking
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caminemos Juntas App (Experimental): Participants use the Caminemos app.
  Interventions: Other: Caminemos Juntas App
- World Walking App (Active Comparator): Participants use the World of Walking App.
  Interventions: Other: World Walking App

INTERVENTIONS:
Other: Caminemos Juntas App — A tailored mobile app that encourages Latinas and Hispanic women to walk together using location-based services.
  Arms: Caminemos Juntas App
Other: World Walking App — A mobile app that encourages users to walk.
  Arms: World Walking App

SUMMARY:
Despite numerous interventions designed to increase physical activity, few are specifically tailored to Latinas, a population where higher rates of obesity, diabetes, and other chronic diseases are present. This proposed smartphone app, ¡Caminemos Juntas!, will use location-based services to connect Latinas with one another in order to improve walking habits by increasing social support and decreasing perceived barriers, both of which are known to play a role in physical activity behaviors. Through a randomized comparative-effectiveness trial, this Phase II project will test the effectiveness of a smartphone application for improving physical activity among Latinas when providing them with real-time opportunities to connect socially with the goal of walking.

DETAILED DESCRIPTION:
Health disparities are high among Latinas. They are more likely to be overweight, diagnosed with diabetes, and physically inactive compared to their non-Hispanic White counterparts. Thus, interventions that target improving health access and ameliorating chronic diseases among Latinas are of high public health importance. Available data suggest that community-focused interventions produce improvements in physical activity (PA) and are well-received by Latinas especially when social and physical environments are considered (e.g., social support, safe walking areas, etc.). Research suggests that Latinos respond favorably to technological-based health interventions. Thus, health promotion interventions that can address Latinos' preferences regarding their physical and social environments while utilizing a preferred technology source (e.g., smartphone) could prove highly successful. In a Phase I SBIR, our team developed ¡Caminemos Juntas!, an innovative mobile phone app using Location-based Services (LBS) to connect women within geographically proximal neighborhoods as a way to provide social support for increased walking behaviors. Specifically, we (a) gathered feedback from an Expert Advisory Board (EAB) to help plan and assess the feasibility of creating the app; (b) built connections and gathered input from Latina community leaders to assist in the conceptual development of the app through a Community Advisory Board (CAB); (c) conducted an online survey of a national sample of Latinas on their smartphone usage for health promotion, and interest in social networking and LBS technology features; (d) conducted iterative focus groups with Latinas to guide development of app content, design, and aesthetics to fully develop a functioning prototype; (e) conducted field usability testing with Latinas to test the app's accuracy to establish users' location and connect users through the ¡Caminemos Juntas! system and users' use and satisfaction with the app; and (f) developed a specifications document to outline the Phase II development plan. The results of the Phase I activities provided strong support for this Phase II SBIR application. The proposed Phase II project will (1) develop a full-scale, fully programmed ¡Caminemos Juntas! app; (2) determine whether the ¡Caminemos Juntas! app can be translated and adapted to a new community environment; (3) test the performance, usage, and usability of the full-scale, fully-programmed app; and (4) evaluate whether ¡Caminemos Juntas! increases physical activity, social support for exercise, and quality of life (QOL) in Latinas. ¡Caminemos Juntas! will be evaluated in a randomized comparative-effectiveness trial (n=200) with Latinas age 18-55 in the Denver, CO and San Jose, CA areas. Overall, the proposed project has the potential to significantly impact Latinas' health by providing them with real-time opportunities to connect socially with the goal of walking. ¡Caminemos Juntas! will be the first app that use geo-location technology dedicated to walking with a social emphasis, for any population.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 69 years, identify as Hispanic or Latina, identify as a woman, able to read and speak either English or Spanish, own a smartphone, not pregnant, consent to participate

Exclusion Criteria:

* Not between the ages of 18 and 69 years, not identify as Hispanic or Latina, not identify as a woman, unable to read or speak Spanish or English, pregnant, not own a smartphone.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PhD, Principal Investigator — Senior Scientist
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Klein Buendel, Inc., Golden, Colorado

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caminemos Juntas App | World Walking App
Started | 38 | 40
Completed | 38 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caminemos Juntas App | World Walking App | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 39 | 75
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 44.26 [18 to 67] | 43.97 [20 to 67] | 44.05 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 40 | 78
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Latino women, ages 18-69 years, were recruited from the Bay area of California and Denver, Colorado (N= 78).
  participants
    United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity at 4 Weeks
Description: The Community Healthy Activities Model Program for Seniors (CHAMPS) is a 41-item PA questionnaire that measures self-reported minutes-per-week of PA calculated as total weekly caloric expenditure for all PA. It was developed for underactive populations and validated among older adults. However, CHAMPS has been used with younger and racially/ethnically diverse populations; it is sensitive to change specifically in Latino and other populations including ones younger than senior age. The CHAMPS asks about activities undertaken for exercise, daily activities that are physical in nature, and physically active recreational activities during "a typical week in the past 4 weeks."
Time Frame: 0 weeks and 4 weeks
Population: Participants with available data at 4 weeks were analyzed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: kilocalories/kg/hour
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 34 | 35
kilocalories/kg/hour | 43.21 (32.87) | 36.76 (29.93)

2. Primary Outcome: Change in Physical Activity at 8 Weeks
Description: The Community Healthy Activities Model Program for Seniors (CHAMPS) is a 41-item physical questionnaire that measures self-reported minutes-per-week of physical activity calculated as total weekly caloric expenditure in all physical activity. Hours and minutes per week were assessed for different types of physical activity. Using body weight and minutes of physical activity (by type), total caloric expenditure was calculated. Data is presented as a T-score with higher values (positive) indicating more calories expended at 8 weeks compared to baseline. Range = 2.5-145.2 kilocalories/kg/hr in the World Walking App condition; range = 6.9-120.1 kilocalories/kg/hr in the Caminemos condition. This measure was administered at 8 weeks to measure changes in physical activity.
Time Frame: Mean change between 0 and 8 week
Population: Participants with available data at 8 weeks were analyzed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: kilocalories/kg/hour
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 37 | 39
kilocalories/kg/hour | 38.07 (25.7) | 30.07 (32.55)

3. Secondary Outcome: Perceived Receipt of Social Support for Exercise at 4 Weeks
Description: The Social Support for Exercise Survey is a 10-item self-report measure that assesses perceived receipt of social support for exercise, i.e., how often their friends or family members (separately rated) encouraged their exercise behaviors during the previous 3 month. Each question uses a likert-type scale ("1/none, 2/rarely, 3/a few times, 4/often, 5/very often") with higher mean score indicating more support from family and friends. Minimum mean score for the scale = 10; maximum mean score = 50.
Time Frame: 4 weeks
Population: Participants with available data at 4 weeks were analyzed for this Secondary Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 34 | 35
units on a scale
  Family | 23.41 (10.93) | 21.14 (10.09)
  Friends | 20.15 (10.14) | 20.86 (9.86)

4. Secondary Outcome: Perceived Receipt of Social Support for Exercise at 8 Weeks
Description: as for outcome 3
Time Frame: 8 weeks
Population: Participants with available data at 8 weeks were analyzed for this Secondary Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 37 | 39
units on a scale
  Family | 20.65 (10.48) | 20.82 (9.56)
  Friends | 17.97 (8.85) | 20.31 (9.50)

5. Secondary Outcome: Functional Health and Well-being at 4 Weeks
Description: The 12-Item Short Form Health Survey (SF-12) is a 12-item questionnaire that measures functional health and well-being (i.e., health-related quality of life; HRQOL). Answer scales include likert-type scales and dichotomous answer choices. The validated scoring for SF-12 was used; scoring is done by linear transformation with the mean score in the general US population being set to 50. Mean scores above 50 indicate better than average self-reported health. Range = 30.7-61.3 units in the physical component in Caminemos condition; range = 28.2-62.2 units in the physical component in the World Walking App condition. For the mental component, range = 14.8-60.7 in Caminemos condition; range = 18.9-62.9 in the World Walking App. Raw scores are provided.
Time Frame: 4 weeks
Population: Participants with available data at 4 weeks were analyzed for this Secondary Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 34 | 35
units on a scale
  Physical Component | 51.33 (7.72) | 50.00 (6.49)
  Mental Component | 47.57 (10.83) | 48.16 (10.90)

6. Secondary Outcome: Functional Health and Well-being at 8 Weeks
Description: The 12-Item Short Form Health Survey (SF-12) is a 12-item questionnaire that measures functional health and well-being (i.e., health-related quality of life; HRQOL). Answer scales include likert-type scales and dichotomous answer choices. The validated scoring for SF-12 was used; scoring is done by linear transformation with the mean score in the general US population being set to 50. Mean scores above 50 indicate better than average self-reported health. Range = 32.0-61.6 units in the physical component in Caminemos condition; range = 32.4-59.2 units in the physical component in the World Walking App condition. For the mental component, range = 28.0-60.8 in Caminemos condition; range = 22.3-60.8 in the World Walking App. Raw scores are provided.
Time Frame: 8 weeks
Population: Participants with available data at 8 weeks were analyzed for this Secondary Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 37 | 39
units on a scale
  Physical Component | 50.07 (7.68) | 50.87 (5.97)
  Mental Component | 49.95 (10.02) | 49.19 (11.01)

7. Secondary Outcome: System Usability Scale (SUS)
Description: Ten likert-type questions assessing user-friendliness of technology. Each question has five answer options that range from 1="Strongly Disagree" to 5="Strongly Agree". Scores range from 0-100. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. A score above 68 is considered above average. Higher scores indicate a more usable technology compared to lower. Raw scores are presented. Range = 20-100 for Caminemos; range = 15-95 for World Walking App. All scores averaged.
Time Frame: 8 weeks
Population: Participants with available data at 8 weeks were analyzed for this Secondary Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caminemos Juntas App | World Walking App
Number analyzed (Participants) | 37 | 39
score on a scale | 60.95 (19.68) | 60.13 (22.09)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Behavioral study did not pose risk for adverse events.
Arm/Group | Caminemos Juntas App | World Walking App
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03854916/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03854916/ICF_001.pdf